CLINICAL TRIAL: NCT06016543
Title: Role of OMT in the Management of the Persistent Post-COVID-19 Symptoms - A Pilot Prospective Cohort Study
Brief Title: Role of OMT in the Management of the Persistent Post-COVID-19 Symptoms
Acronym: ROMPS
Status: Completed | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Other Study IDs: ROMPS-Pilot
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: osteopathic manipulative treatment; long COVID; post-COVID conditions; post-acute sequelae of SARS-CoV-2 infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: osteopathic manipulative treatment (OMT) — Osteopathic manipulative treatment provided at the discretion of the treating physician and based on the patient's response to previous treatments.

SUMMARY:
The goal of this observational study is to determine the feasibility of conducting a large-scale study on the effect of using osteopathic manipulative treatment (OMT) to treat patients with post-COVID-19 symptoms. The main questions it aims to answer are:

1. Is it feasible to conduct a large-scale study of the effect of OMT on patients with post-COVID-19 symptoms (based on how many patients agree to participate and how many complete the study)?
2. How much change in patients' post-COVID-19 symptom severity, quality of life, and ability to return to work can we expect to see following OMT?

Participants will receive OMT as directed by their physician and complete questionnaires after every other OMT session.

1. Participants will complete questionnaires about their post-COVID-19 symptoms, quality of life, ability to return to work, and adverse events they experienced 3 days after every other OMT session.
2. Participants will be sent links to the questionnaires for 4 months or when their symptoms resolve, whichever comes first.
3. Additionally, participants will complete a follow-up questionnaire 2 months after they stop receiving OMT for their post-COVID-19 symptoms or 6 months after enrollment in the study, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* at least one symptom of post-COVID-19 (eg, fatigue, dyspnea, anosmia, arthralgia, headache, sleep disturbances, anxiety/depression, or other problems related to mental health) which was new after diagnosis with COVID-19 and has persisted for at least 4 weeks after diagnosis

Exclusion Criteria:

* unable to speak, read, and write in English
* not mentally competent to give informed consent
* inability to complete surveys/questionnaires online

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of clinics in the United States where members of the practice-based research network, DO-Touch.NET, practice osteopathic manipulative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Patient recruitment rate (feasibility) | Through study completion, an average of 1 year
  Proportion of patients who enroll in the study out of the number of patients who were eligible for and invited to enroll in the study.
Data completion rate (feasibility) | Through study completion, an average of 1 year
  Proportions of participants and physicians who complete all their questionnaires.

SECONDARY OUTCOMES:
Neurocognitive and psychological symptoms | 3 days after every other OMT session for up to 4 months after enrollment and 2 months after the participant's final OMT session
  Measured using the Rivermead Post Concussion Symptoms Questionnaire
Physical symptoms | 3 days after every other OMT session for up to 4 months after enrollment and 2 months after the participant's final OMT session
  Measured using the Long COVID-Household Pulse Survey
Global health | 3 days after every other OMT session for up to 4 months after enrollment and 2 months after the participant's final OMT session
  Measured using the PROMIS SF v1.2 Global Health scale
Return to work | 3 days after every other OMT session for up to 4 months after enrollment and 2 months after the participant's final OMT session
  For participants who were employed prior to COVID-19, their current working status will be assessed on a 4-point scale (1. returned to full-time work without restrictions, 2. returned to full-time work but with modified job duties, 3) returned to work but with reduced working hours, 4. have not been able to return to work.

OTHER OUTCOMES:
Severity of potential adverse events from OMT | 3 days after every other OMT session for up to 4 months after enrollment
  Measured by comparing the severity of potential adverse events from OMT during the 3 days following OMT to the severity during the week before OMT.

CONTACTS AND LOCATIONS:
Overall Officials: Brian F Degenhardt, DO, Principal Investigator — A.T. Still University of Health Sciences
Locations (1):
- Osteopathic Manipulative Medicine Gutensohn Clinic, Kirksville, Missouri, United States

IPD SHARING:
Plan to Share IPD: No